CLINICAL TRIAL: NCT01208792
Title: Auto-immunity and Prognosis of Pulmonary Arterial Hypertension
Brief Title: Auto-immunity and Pulmonary Arterial Hypertension
Acronym: Auto-HTAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: P071209
Record Dates: First submitted 2010-07-12; First posted 2010-09-24 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension; HIV Infection; Congenital Heart Defect; Systemic Sclerosis; Connective Tissue Disease
Keywords: Auto antibodies; Target antigens; 2D-immunoblot; Reactive oxygen species; Pulmonary arterial hypertension; Systemic sclerosis; Human immunodeficiency virus infection; Porto pulmonary hypertension; Congenital heart defect; Systemic lupus erythematosus; Mixed connective tissue disease; Sjögren's syndrome
MeSH Terms: conditions — Pulmonary Arterial Hypertension; HIV Infections; Heart Defects, Congenital; Scleroderma, Systemic; Connective Tissue Diseases; Acquired Immunodeficiency Syndrome; Lupus Erythematosus, Systemic; Mixed Connective Tissue Disease; Sjogren's Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Disease group (Experimental): Two hundred patients with PAH will be included: 50 patients with idiopathic PAH (iPAH), 20 with PAH associated with HIV infection, 20 with porto-pulmonary hypertension, 20 with PAH secondary to congenital heart disorders, 40 with SSc, 20 with SLE, 20 with MCTD and 10 with a PAH associated with a Sjögren's syndrome. Two hundred patients without PAH will also be included: 80 patients with SSc and 20 in each of the following groups: HIV infection, porto-pulmonary hypertension, SLE, congenital heart disorders, MCTD and with Sjögren's syndrome.
  Interventions: Procedure: skin biopsy; Other: Blood Sample
- Control group 1 (Other): Two hundred healthy blood donors age and sex-matched with patients with PAH, will be included as controls.
  Interventions: Other: Blood Sample
- Control group 2 (Other): Twenty patients with proximal chronic thromboembolic pulmonary hypertension (CTPH) will also be included in a control arm of the study.
  Interventions: Other: Blood Sample

INTERVENTIONS:
Procedure: skin biopsy — The biopsy site (usually the forearm) will be first cleaned, and then anesthetized with pain relieving (spray, cream, or injection). The skin is then sampled using a punch that takes a core (a small cylindrical fragment of tissue from the area of interest
  Arms: Disease group
Other: Blood Sample — a blood sample will be collected

SUMMARY:
The investigators have recently evidenced the presence of antibodies to endothelial cells and fibroblasts in patients with idiopathic or SSc-associated PAH. The investigators also have identified several target antigens of anti-fibroblasts antibodies.

The objective of this study is to further investigate for the presence of antibodies to endothelial cells and fibroblasts in patients and characterize the antigen specificity of autoantibodies in patients with different types of non idiopathic and non SSc-associated PAH, such as PAH associated with HIV infection, porto-pulmonary hypertension, congenital heart diseases, systemic lupus erythematosus, mixed connective tissue disease and Sjögren's syndrome

DETAILED DESCRIPTION:
Two hundred and fifty patients with PAH will be included: 65 patients with idiopathic PAH (iPAH), 20 with PAH associated with HIV infection, 20 with porto-pulmonary hypertension, 20 with PAH secondary to congenital heart disorders, 40 with SSc, 20 with SLE, 20 with MCTD and 10 with a PAH associated with a Sjögren's syndrome.

Two hundred patients without PAH will also be included: 80 patients with SSc and 20 in each of the following groups: HIV infection, porto-pulmonary hypertension, SLE, congenital heart disorders, MCTD and with Sjögren's syndrome.

Twenty patients with proximal chronic thromboembolic pulmonary hypertension (CTPH) will also be included in a control arm of the study.

Two hundred and fifty healthy blood donors age and sex-matched with patients with PAH, will be included as controls.

By using 2D-immunoblotting techniques, we will evidence IgG antibodies to fibroblasts, EC, vascular smooth muscle cells (SMC) in multiple groups of patients and we will characterize target antigens of these autoantibodies. We will also assess the production of ROS: nitric oxide (NO), hydrogen peroxide (H2O2) and the effect of the whole serum (and the IgG particularly) on in VITRO proliferation of EC, fibroblasts and vascular SMC. For sera that will induce the production of ROS, we will study the effect of different vasodilatator (prostacycline, endothelin receptor antagonist, type 5 phosphodiesterase inhibitors) and anti-oxidant therapies.

Expected results We will characterize target antigens of autoantibodies of patients with non-idiopathic and non SSc-associated PAH. We will compare these target to those previously identified in idiopathic or SSc-associated PAH. We will then, distinguish subpopulations of PAH patients whose serum or purified IgG (possibly specific for a given antigen) are able to induce ROS production or cell proliferation. For the population of ROS-producer patients, we will correlate the clinical response to vasodilatator therapy to results of in VITRO inhibition experiments with vasodilatators and anti-oxidant molecules.

Perspectives The characterization of target antigens of EC, fibroblasts and vascular SMC specifically

ELIGIBILITY:
Inclusion Criteria:

age over 18

* for PAH patients: pre-capillary PAH evidenced by right-heart catheterization
* no associated systemic disease for idiopathic PAH patients
* for HIV patients, HIV1 infection confirmed by ELISA and western blot
* for patients with porto pulmonary hypertension: evidence by endoscopy of esophageal varices, confirmation of hepatic venous pressure gradient over 5 mmHg by catheterization of the hepatic veins
* for patients with congenital heart defect: evidence by imaging of atrial or ventricular septal defect, or patent ductus arterious and confirmed by heart catheterization
* patients with SSc will fulfill the American College of Rheumatology (ACR) and the LEROY and MEDSGER criteria
* patients with MCTD will fulfill the criteria for MCTD
* patients with SLE will fulfill the updated and revised ACR criteria
* patients with Sjögren's syndrome will fulfill the American-European consensus group criteria
* patients with chronic thromboembolic pulmonary hypertension: Lung scintiscan showing segmental mismatched perfusion defects and confirmation by angiography of the occlusion and the chance of success of endarterectomy according to the location of disease
* Signed written informed consent
* Patients with health insurance

Exclusion Criteria:

* age under 18
* pregnant women
* absence of written informed consent
* associated malignant tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 629 (Actual)
Dates: Start 2010-06-15 (Actual); Primary Completion 2014-07-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Immunological markers of prognosis interest in pulmonary arterial hypertension (PAH) | one year

SECONDARY OUTCOMES:
Target antigens of autoantibodies | one year
  To characterize target antigens of autoantibodies in non-idiopathic and non-SSc associated PAH and to compare these target antigens to those recognized by autoantibodies directed at endothelial cells, fibroblasts and vascular smooth muscle cells in patients with idiopathic and SSc-associated PAH;
Subpopulations of patients with PAH whose serum is able to induce the production of reactive oxygen species (ROS) | one year
  * To study and characterize subpopulations of patients with PAH whose serum is able to induce the production of reactive oxygen species (ROS) and/or cell proliferation.
  * In patients in whom the whole serum induces cell proliferation and ROS production in cell cultures, to correlate the results of inhibition experiments in vivo in the presence of vasodilators used in the treatment of PAH and clinical response to these vasodilators

CONTACTS AND LOCATIONS:
Overall Officials: Luc Mouthon, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (3):
- France (3):
  - Pneumology Department, Antoine Béclère Hospital, Clamart
  - Internal Medicine Department, Claude Huriez Hospital, Lille
  - Internal Medicine Department, Cochin Hospital, Paris